CLINICAL TRIAL: NCT00436826
Title: A Phase II, Multicenter, Randomized, Double Blind, Placebo Controlled, Safety, Tolerability and Efficacy Study of Add-on Cladribine Tablet Therapy With Interferon-beta (IFN-β) Treatment in Multiple Sclerosis Subjects With Active Disease
Brief Title: A Phase 2 Study of Cladribine Add-on to Interferon-beta (IFN-beta) Therapy in Multiple Sclerosis (MS) Subjects With Active Disease (ONWARD)
Acronym: ONWARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26593; 2006-003366-33 (EudraCT Number)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing forms; Interferon-beta therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine; Interferon-beta; Interferon beta-1a; Interferon beta-1b

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Cladribine 3.5 mg/kg, IFN-beta (DB period) (Experimental): Participants received cladribine tablets orally as cumulative dose of 0.875 mg/kg over a course of 4-5 consecutive days at Week 1, 5, 48, and 52 resulting in total cladribine dose of 3.5 milligram per kilogram (mg/kg) along with interferon (IFN)-beta therapy (Rebif® new formulation [RNF] 44 mcg three times a week, subcutaneously; Avonex® 30 microgram (mcg) every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) during the Double blind period (DBP) of 96 weeks.
  Interventions: Drug: Cladribine; Drug: Interferon-beta (IFN-beta)
- Placebo, IFN-beta (DB period) (Placebo Comparator): Participants received matching placebo tablets orally over a course of 4-5 consecutive days at Week 1, 5, 48, and 52 along with IFN-beta therapy (RNF 44 mcg three times a week, subcutaneously; Avonex® 30 mcg every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) during the DB period of 96 weeks.
  Interventions: Drug: Placebo; Drug: Interferon-beta (IFN-beta)
- Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) (Experimental): Participants who received cladribine 3.5 mg/kg initially and completed DB period entered in the open label (OL) extension (Ext.) period. In OL Ext. period, participant who met the eligibility criteria received OL oral cladribine 3.5 mg/kg over maximum of 48 weeks along with IFN-beta therapy (RNF 44 mcg three times a week, subcutaneously; Avonex® 30 mcg every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) up to 48 weeks.
  Interventions: Drug: Cladribine; Drug: Interferon-beta (IFN-beta)
- Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) (Placebo Comparator): Participants who received placebo initially and completed DB period entered in the OL Ext. period. In OL Ext. period, participant who met the eligibility criteria received OL oral cladribine 3.5 mg/kg over maximum of 48 weeks along with IFN-beta therapy (RNF 44 mcg three times a week, subcutaneously; Avonex® 30 mcg every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) up to 48 weeks.
  Interventions: Drug: Cladribine; Drug: Placebo; Drug: Interferon-beta (IFN-beta)
- Cladribine 3.5 mg/kg, IFN-beta (Safety follow up) (Experimental): Participants who received cladribine 3.5 mg/kg initially and completed DB period entered in the OL ext. safety follow up period. In this period, participants who did not meet eligibility criteria received only IFN-beta therapy (RNF 44 mcg three times a week, subcutaneously; Avonex® 30 mcg every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) up to 48 weeks.
  Interventions: Drug: Cladribine; Drug: Interferon-beta (IFN-beta)
- Placebo, IFN-beta (Safety follow up) (Placebo Comparator): Participants who received placebo initially and completed DB period entered in the OL ext. safety follow up period. In this period, participants who did not meet eligibility criteria received only IFN-beta therapy (RNF 44 mcg three times a week, subcutaneously; Avonex® 30 mcg every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) up to 48 weeks.
  Interventions: Drug: Placebo; Drug: Interferon-beta (IFN-beta)

INTERVENTIONS:
Drug: Cladribine — Participants were administered with cladribine tablets orally as cumulative dose.
  Arms: Cladribine 3.5 mg/kg, IFN-beta (DB period); Cladribine 3.5 mg/kg, IFN-beta (Safety follow up); Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext); Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Drug: Placebo — Participants were administered with placebo orally.
  Arms: Placebo, IFN-beta (DB period); Placebo, IFN-beta (Safety follow up); Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Drug: Interferon-beta (IFN-beta) — Participants received IFN-beta therapy (Rebif® new formulation [RNF] 44 microgram [mcg] three times a week, subcutaneously; Avonex® 30 mcg every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) during both DB period of 96 weeks and OL extension period of 48 weeks.
  Other Names: Avonex®; Betaseron®; RNF

SUMMARY:
The goal of this study was to evaluate the safety, tolerability and effectiveness of oral cladribine when taken in combination with Interferon-beta (IFN-beta) therapy for the treatment of multiple sclerosis (MS).

This study randomized around 200 participants from approximately 50 sites located world-wide, who have experienced at least one relapse while taking IFN-beta therapy within 48 weeks prior to Screening, irrespective of disability progression. Secondary progressive multiple sclerosis (SPMS) participants, who were still experiencing relapses, and participants who have received disease modifying drugs (DMDs), other than IFN-beta therapy, during their MS treatment history, but were currently on IFN-beta therapy and have experienced active MS symptoms (at least 1 relapse) during the 48 weeks prior to Screening, were enrolled.

Participants were randomized in a 2:1 fashion to receive up to 4 cycles of oral cladribine or matching placebo in combination with IFN-beta therapy. Participants who completed the double-blind portion of the study were invited to participate in an open-label extension phase of matching study design.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, 18 to 65 years of age (inclusive)
* Weigh between 40 to 120 kilogram (kg), (inclusive)
* Have definite MS, as confirmed by the revised McDonald criteria 2005, and have relapsing forms of MS, such as relapsing-remitting multiple sclerosis (RRMS) or SPMS with superimposed relapses
* Have experienced at least one relapse within 48 weeks prior to Screening, while receiving IFN-beta treatments (Rebif® 44mcg three times a week, subcutaneously; Avonex®30 mcg every week, intramuscular; or Betaseron® 250 mcg every other day, subcutaneously)
* Have a minimum time on IFN-beta therapy of 48-consecutive weeks prior to Screening. Participants who switched from one IFN-beta therapy to another in the 48 weeks preceding Screening may be entered into the study if they have been on a stable regimen of their current IFN-beta therapy for a minimum of 3 months prior to Screening
* Be clinically stable (other than MS relapse) during the 28 days preceding Screening
* The following hematological parameters must be normal (as defined below, inclusively) within 28 days of first dosing of blinded study medication at study day 1 (SD 1)

  * Hemoglobin=11.6 to 16.2 gram per deciliter (g/dL)
  * Leukocytes (total white blood cells [WBC])=4.1 to 12.3*10^3 per microliter (/UL)
  * Absolute lymphocytes count (ALC)= 1.02 to 3.36*10^3/UL
  * Absolute neutrophil count (ANC)=2.03 to 8.36*10^3/UL
  * Platelet count=140 to 450*10^3/UL
* Have no medical history or evidence of latent tuberculosis infection (LTBI) or active tubercular disease (TB), as evidenced by TB skin test or chest X-ray
* Have an expanded disability status scale (EDSS) from 1.0-5.5, inclusive
* Have no prior exposure to immunosuppressive or cytotoxic agents (with the exception of steroids for MS flare management, or intravenous immunoglobulin-G [IVIG] after allowed wash-out periods
* If female, must:

  * be neither pregnant nor breast-feeding, nor attempting to conceive, and
  * use a highly effective method of contraception throughout the entire duration of the study and for 6 months (6 menstrual cycles) following completion of the last dose of study medication. A highly effective method of contraception is defined as one which result in a low failure rate (that is, less than 1 percent per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or a vasectomized partner. For the purpose of this trial, women of childbearing potential are defined as: All female participants after puberty unless they are post-menopausal for at least 2 years, or are surgically sterile
* If male, must be willing to use contraception to avoid pregnancies throughout the entire duration of the study and for 90 days following the last dose of study medication
* Be willing and able to comply with study procedures for the duration of the study
* Have not met any of the exclusion criteria outlined below; and
* Have voluntarily provided written informed consent, including, for United states of America (USA), participant authorization under Health Insurance Portability and Accountability Act (HIPAA), prior to any study-related procedure that is not part of normal medical care, and with the understanding that the participant may withdraw consent at any time without prejudice to future medical care
* Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* Has primary progressive multiple sclerosis (PPMS) or SPMS without relapses forms
* Has prior or current malignancy other than medically documented complete excision of basal cell skin cancer no less than 5 years prior to Screening
* Has a history of chronic or clinically significant hematological abnormalities
* Prior use of cladribine, fingolimod, teriflunimide, laquinimod, mitoxantrone, campath-1h, cyclophosphamide, azathioprine, methotrexate, daclizumab, natalizumab, lymphoid irradiation, bone marrow transplantation or myelosuppressive/cytotoxic therapy
* Use of cytokine or anti-cytokine therapy or plasmapheresis within 3 months prior to SD 1
* Treatment with IVIG within 30 days of Screening
* Treatment with oral or parenteral corticosteroids 30 days of Screening
* Treatment with adrenocorticotropic hormone within 28 days prior to SD 1
* Use of any investigational drug (other than Rebif® New Formulation [RNF], Avonex® or Betaferon®) or experimental procedure within 6 months prior to SD 1
* Has inadequate liver function, defined by a total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase greater than 2.5 times the upper limit of the normal values
* Suffers from major medical illness such as cardiac, endocrinologic, hepatic, immunologic (other than MS), metabolic, renal, pulmonary, gastrointestinal, dermatologic, or other major disease that would preclude the administration of oral cladribine
* Suffers from major psychiatric illness (including history of, or current, severe depressive disorders and/or suicidal ideation) that in the opinion of the investigator creates undue risk to the participant or could affect compliance with the study protocol
* Has history of active or chronic infectious disease or any disease which compromises immune function (for example, human immunodeficiency virus [HIV]+, human T-lymphotropic virus [HTLV-1], Lyme disease, LTBI or TB)
* Has an allergy or hypersensitivity to gadolinium, to cladribine or any of its excipients, or IFN-beta or any of its excipient(s)
* Has any renal condition that would preclude the administration of gadolinium (for example, acute or chronic severe renal insufficiency [glomerular filtration rate less than 30 milliliter per minute {mL/min} per 1.73 square meter {m^2}])
* Has a positive stool hemoccult test at Screening
* Has a history of seizures not adequately controlled by treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2006-11-30 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2012-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (39):
- United States (21):
  - Research Site, Cullman, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Boulder, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Peoria, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Newark, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Burlington, Vermont
- Italy (4):
  - Research Site, Fidenza
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Rome
- Russia (7):
  - Research Site, Arkhangelsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Smolensk
- Spain (7):
  - Research Site, Alicante
  - Research site, Barcelona
  - Research Site, Bilbao
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago
  - Research Site, Seville

REFERENCES:
- [Derived] Giovannoni G, Galazka A, Schick R, Leist T, Comi G, Montalban X, Damian D, Dangond F, Cook S. Pregnancy Outcomes During the Clinical Development Program of Cladribine in Multiple Sclerosis: An Integrated Analysis of Safety. Drug Saf. 2020 Jul;43(7):635-643. doi: 10.1007/s40264-020-00948-x. PMID 32447743
- [Derived] Montalban X, Leist TP, Cohen BA, Moses H, Campbell J, Hicking C, Dangond F. Cladribine tablets added to IFN-beta in active relapsing MS: The ONWARD study. Neurol Neuroimmunol Neuroinflamm. 2018 Jul 11;5(5):e477. doi: 10.1212/NXI.0000000000000477. eCollection 2018 Sep. PMID 30027104
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=26593
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initially 42 participants randomized under original protocol but enrollment terminated because of hematological toxicities. Protocol amendment 1 and 2 were implemented and enrolled 172 participants. Protocol amendment 5 was generated, resulting in discontinuation of Cladribine and reduction of Extension period and Safety Follow up to 48 weeks.
Period: Double Blind Period (DBP)
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period) | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) | Placebo, IFN-beta (Safety Follow up)
Started | 124 | 48 | 0 | 0 | 0 | 0
Completed | 111 | 37 | 0 | 0 | 0 | 0
Not Completed | 13 | 11 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 10 | 11 | 0 | 0 | 0 | 0
Period: Ext. Period (With Cladribine Treatment)
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period) | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) | Placebo, IFN-beta (Safety Follow up)
Started | 0 | 0 | 47 | 28 | 0 | 0
Completed | 0 | 0 | 1 | 2 | 0 | 0
Not Completed | 0 | 0 | 46 | 26 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other un-specified | 0 | 0 | 46 | 25 | 0 | 0
Period: Ext. Period (No Cladribine Treatment)
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period) | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) | Placebo, IFN-beta (Safety Follow up)
Started | 0 | 0 | 0 | 0 | 52 | 7
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 51 | 7
Not completed — Sponsor's decision to terminate study | 0 | 0 | 0 | 0 | 51 | 7

BASELINE CHARACTERISTICS:
Groups:
- Cladribine 3.5 mg/kg, IFN-beta: Participants received cladribine tablets orally as cumulative dose of 0.875 milligram per kilogram (mg/kg) over a course of 4-5 consecutive days at Week 1, 5, 48, and 52 resulting in total cladribine dose of 3.5 mg/kg along with IFN-beta therapy (Rebif® new formulation [RNF] 44 microgram [mcg] three times a week, subcutaneously; Avonex® 30 mcg every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) during the double blind (DB) period of 96 weeks. After completing DB period, participants entered in OL extension period. In OL extension period, participant who met eligibility criteria received OL oral cladribine 3.5 mg/kg and participants who did not meet the eligibility criteria received IFN-beta only and were followed for safety only.
- Placebo, IFN-beta: Participants received matching placebo tablets orally over a course of 4-5 consecutive days at Week 1, 5, 48, and 52 along with IFN-beta therapy (RNF 44 mcg three times a week, subcutaneously; Avonex® 30 mcg every week, intramuscularly; or Betaseron® 250 mcg every other day, subcutaneously) during the double blind (DB) period of 96 weeks. After completing DB period, participants entered in OL extension period. In OL extension period, participant who met eligibility criteria received OL oral cladribine 3.5 mg/kg and participants participants who did not meet the eligibility criteria received IFN-beta only and were followed for safety only.
- Total: Total of all reporting groups
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta | Placebo, IFN-beta | Total
Number analyzed (Participants) | 124 | 48 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10.2) | 40.1 (10.3) | 38.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 36 | 120
  Male | 40 | 12 | 52
Time (years) from first attack to study Day 1 [Mean (Standard Deviation); unit: years] | 9.98 (7.24) | 10.83 (7.98) | 10.22 (7.44)
Expanded disability status scale (EDSS) score [Mean (Standard Deviation); unit: unit on scale] — Expanded disability status scale (EDSS) assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated.
  unit on scale | 2.9 (1.2) | 3.0 (1.2) | 2.9 (1.2)
Number of Gadolinium-enhanced lesions [Mean (Standard Deviation); unit: lesions] | 1.1 (4.0) | 0.6 (1.2) | 0.9 (3.4)
Number of Time constant 1 (T1) hypointense lesions [Mean (Standard Deviation); unit: lesions] | 9.0 (9.2) | 9.3 (9.9) | 9.1 (9.3)
T1 Gd+ volume [Mean (Standard Deviation); unit: cubic millimetre (mm^3)] | 150.3 (592.2) | 99.4 (210.0) | 136.1 (514.5)
T2 lesions volume [Mean (Standard Deviation); unit: mm^3] | 10791.2 (11298.0) | 13669.1 (16605.2) | 11596.3 (13013.5)

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Period: Percentage of Participants With Grade 3 or 4 (Common Terminology Criteria for Adverse Events [CTCAE] v 4.0) Hematological or Liver Toxicity
Description: Percentage of participants with Grade 3 or 4 CTCAE v 4.0 toxicity on the following hematology and liver function parameters were reported: lymphocytes, cluster of differentiation 4 (CD4) cell, neutrophils, white blood cells, hemoglobin, Alanine transaminase (ALT), Aspartate transaminase (AST), Platelets and Bilirubin. According to CTCAE v 4.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death.
Time Frame: Baseline up to Week 96
Population: Safety population: all randomized participants who received at least 1 dose of study drug in DBP and had follow-up safety data.
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 124 | 48
Percentage of participants
  Grade 3 or 4 Lymphocyte toxicity | 63.71 | 2.08
  Grade 3 or 4 Hemoglobin toxicity | 2.42 | 0.00
  Grade 3 or 4 White Blood Cell toxicity | 10.48 | 0.00
  Grade 3 or 4 Neutrophil toxicity | 12.10 | 2.08
  Grade 3 or 4 CD4+ toxicity | 50.81 | 2.08
  Grade 3 or 4 AST toxicity | 0.81 | 0.00
  Grade 3 or 4 ALT toxicity | 0.81 | 2.08
  Grade 3 or 4 Platelet toxicity | 0.00 | 0.00
  Grade 3 or 4 Bilirubin toxicity | 0.00 | 0.00

2. Primary Outcome: Double Blind Period: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) in Infections and Infestations System Organ Class (SOC)
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration.TEAEs were entered in infections and infestations SOC as per medical dictionary for regulatory activities (MedDRA) version 11.0
Time Frame: Baseline up to Week 96
Population: Safety population included all randomized participants who received at least one dose of study medication in the DBP and had follow-up safety data.
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 124 | 48
Percentage of participants | 61.3 | 54.2

3. Primary Outcome: Double Blind Period: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered. SAE: Any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Week 96
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 124 | 48
Participants
  Participants with TEAEs | 119 | 36
  Participants with Serious TEAEs | 12 | 5

4. Primary Outcome: Double Blind Period: Time to First Grade 3 or 4 Hematological Toxicity or Liver Toxicity
Description: Time to first Grade 3 or 4 hematological toxicity or liver toxicity (lymphocytes, cluster of differentiation 4 (CD4) cell, neutrophils, white blood cells, hemoglobin, Alanine transaminase (ALT), Aspartate transaminase (AST), Platelets and Bilirubin) were estimated using the Kaplan-Meier method. According to CTCAE v 4.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death. 10th and 20th percentiles estimated from Kaplan-Meier survival curve. Due to the small number of events, estimates from Kaplan-Meier survival curves could only be derived for lower percentiles. The median (50th percentile) could not be estimated if less than 50% of the participants had an event during the time of the study. Accordingly, lower percentiles are presented according to the number of events observed.
Time Frame: Baseline up to Week 96
Population: Safety population included all randomized participants who received at least one dose of study medication in the DBP and had follow-up safety data. Here "Number of Participants analyzed"= participants evaluable for this outcome measure and "number analyzed"= participants who were evaluable for specified category.
Measure: Number; unit: Months
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 79 | 2
Months
  10th percentile: Lymphocytes toxicity: number analyzed (Participants) | 79 | 1
  10th percentile: Lymphocytes toxicity | 1.61 | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: Lymphocytes toxicity: number analyzed (Participants) | 79 | 1
  20th percentile: Lymphocytes toxicity | 2.00 | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile:Hemoglobin toxicity: number analyzed (Participants) | 2 | 0
  10th percentile:Hemoglobin toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  20th percentile:Hemoglobin toxicity: number analyzed (Participants) | 2 | 0
  20th percentile:Hemoglobin toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  10th percentile: White Blood Cell toxicity: number analyzed (Participants) | 13 | 0
  10th percentile: White Blood Cell toxicity | 17.74 |
  20th percentile: White Blood Cell toxicity: number analyzed (Participants) | 13 | 0
  20th percentile: White Blood Cell toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  10th percentile: Neutrophil toxicity: number analyzed (Participants) | 15 | 2
  10th percentile: Neutrophil toxicity | 12.55 | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: Neutrophil toxicity: number analyzed (Participants) | 15 | 2
  20th percentile: Neutrophil toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: Platelets toxicity: number analyzed (Participants) | 0 | 0
  20th percentile: Platelets toxicity: number analyzed (Participants) | 0 | 0
  10th percentile: CD4+ count toxicity: number analyzed (Participants) | 63 | 2
  10th percentile: CD4+ count toxicity | 1.87 | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: CD4+ count toxicity: number analyzed (Participants) | 63 | 2
  20th percentile: CD4+ count toxicity | 2.99 | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: AST toxicity: number analyzed (Participants) | 1 | 0
  10th percentile: AST toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  20th percentile: AST toxicity: number analyzed (Participants) | 1 | 0
  20th percentile: AST toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  10th percentile: ALT toxicity: number analyzed (Participants) | 1 | 1
  10th percentile: ALT toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: ALT toxicity: number analyzed (Participants) | 1 | 1
  20th percentile: ALT toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: Bilirubin toxicity: number analyzed (Participants) | 0 | 0
  20th percentile: Bilirubin toxicity: number analyzed (Participants) | 0 | 0

5. Primary Outcome: Double Blind Period: Time to Recovery From Grade 3 or 4 Hematological Toxicity
Description: Time to recovery from grade 3 or 4 hematological were reported: lymphocytes, platelets, neutrophils, white blood cells and hemoglobin. According to CTCAE v 4.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death. Recovery" as "Recovery from a Grade 3 or 4 toxicity is defined as a return to a Grade 0 or 1.
Time Frame: Baseline up to Week 96
Population: Safety population: all randomized participants who received at least 1 dose of study drug in DBP and had follow-up safety data. Here "Number of Participants analyzed"= participants evaluable for this outcome measure and "number analyzed"= participants who had a Grade 3 or 4 abnormality and evaluable at specified category.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 76 | 2
Days
  Hemoglobin: number analyzed (Participants) | 2 | 0
  Hemoglobin | 19.50 (10.61) |
  White Blood Cell: number analyzed (Participants) | 13 | 0
  White Blood Cell | 31.27 (27.69) |
  Neutrophil: number analyzed (Participants) | 15 | 2
  Neutrophil | 41.17 (37.90) | 56.75 (30.76)
  Platelet: number analyzed (Participants) | 0 | 0
  Lymphocyte: number analyzed (Participants) | 76 | 1
  Lymphocyte | 142.53 (109.86) | 28.00

6. Primary Outcome: Double Blind Period: Mean Changes in Lymphocytes, White Blood Cells (WBC), Neutrophils and Platelets Values From Baseline to Week 96
Description: Mean changes in lymphocytes, WBC, neutrophils and platelets from baseline to week 96 were reported.
Time Frame: Baseline, Week 96
Population: Safety population: all randomized participants who received at least 1 dose of study drug in DBP and had follow-up safety data. Here "Number of Participants analyzed"= participants evaluable for this outcome measure and "number analyzed"= participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 102 | 33
10^9 cells per liter
  Lymphocytes: number analyzed (Participants) | 102 | 32
  Lymphocytes | -0.8 (0.5) | 0.0 (0.7)
  Platelet: number analyzed (Participants) | 100 | 33
  Platelet | -29.8 (37.9) | -12.4 (56.9)
  WBC | -1.5 (1.8) | -0.4 (1.6)
  Neutrophils: number analyzed (Participants) | 102 | 32
  Neutrophils | -0.7 (1.6) | -0.4 (1.2)

7. Primary Outcome: Double Blind Period: Maximum Corrected QT Interval (QTc)
Description: Criteria for potential clinical concern in ECG parameters: Maximum corrected QT interval (QTc) in range of 450 to less than 480 millisecond (msec).
Time Frame: Baseline up to Week 96
Population: Safety population included all randomized participants who received at least one dose of study medication in the DB period and had follow-up safety data.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 124 | 48
Milliseconds | 0.4381 (0.0194) | 0.4361 (0.0176)

8. Primary Outcome: Double Blind Period: Mean Change From Baseline in Vital Signs- Systolic and Diastolic Blood Pressure
Description: Mean change from baseline in vital signs- systolic and diastolic blood pressure was reported.
Time Frame: Baseline, Week 96
Population: Safety population included all randomized participants who received at least one dose of study medication in the DB period and had follow-up safety data. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mm*hg)
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 113 | 38
Millimeter of mercury (mm*hg)
  Systolic Blood Pressure | -0.6 (13.2) | 0.0 (13.1)
  Diastolic Blood Pressure | -0.6 (10.1) | -2.2 (8.9)

9. Primary Outcome: Double Blind Period: Mean Change From Baseline in Vital Signs- Pulse Rate
Description: Mean change from baseline in vital signs- Pulse Rate was reported.
Time Frame: Baseline, Week 96
Population: Safety population: all randomized participants who received at least 1 dose of study drug in DBP and had follow-up safety data. Here "Number of Participants analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: beats per minutes
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 112 | 38
beats per minutes | 1.0 (11.6) | 0.4 (9.2)

10. Primary Outcome: Double Blind Period: Mean Change From Baseline in Vital Signs- Weight
Description: Mean change from baseline in vital signs- weight was reported.
Time Frame: Baseline, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 111 | 38
Kilogram | -0.6 (8.0) | -0.4 (5.0)

11. Primary Outcome: Double Blind Period: Mean Change From Baseline in Vital Signs- Temperature
Description: Mean change from baseline in vital signs- temperature was reported.
Time Frame: Baseline, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 112 | 38
Degree celsius | -0.1 (0.3) | -0.1 (0.4)

12. Primary Outcome: Double Blind Period: Mean Change From Baseline in Electrocardiogram (ECG) Parameters- Heart Rate
Description: Mean change from baseline in ECG parameters- Heart Rate was reported.
Time Frame: Baseline, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats per minutes
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 37 | 22
beats per minutes | -3.114 (8.990) | 1.981 (7.857)

13. Primary Outcome: Double Blind Period: Mean Change From Baseline in Electrocardiogram (ECG) Parameters- PR, RR, QRS and OT Interval
Description: Mean change from baseline in ECG parameters- PR, RR, QRS and OT interval was reported.
Time Frame: Baseline, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 37 | 22
milliseconds
  PR Interval | 0.0001 (0.0094) | 0.0033 (0.0108)
  RR Interval | 0.0361 (0.1068) | -0.0272 (0.1175)
  QRS Interval | 0.0028 (0.0060) | 0.0043 (0.0054)
  QT Interval | 0.0135 (0.0214) | 0.0037 (0.0189)

14. Primary Outcome: Double Blind Period: Mean Changes From Baseline in Hemoglobin Level to Week 96
Description: Mean changes in hemoglobin level from baseline to week 96 was reported.
Time Frame: Baseline, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 102 | 33
gram per liter (g/L) | -2.9 (8.1) | -2.5 (10.6)

15. Primary Outcome: Double Blind Period: Mean Changes From Baseline in CD4+ Count, CD8+ Count, and CD19+ to Week 96
Description: Mean changes CD4+ Count, CD8+ Count, and CD19+ from baseline to Week 96 were reported.
Time Frame: Baseline, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 99 | 31
Cells per microliter
  CD4+ | -604.1 (301.3) | 7.1 (344.7)
  CD8+ | -137.8 (178.1) | 23.9 (188.3)
  CD19+ | 22.0 (141.2) | 30.7 (121.5)

16. Primary Outcome: Double Blind Period: Mean Changes From Baseline in Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) to Week 96
Description: Mean changes in ALT and AST from baseline to week 96 were reported.
Time Frame: Baseline, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 102 | 32
Units per liter
  ALT | -3.0 (11.5) | 1.3 (11.5)
  AST | -1.7 (6.9) | 1.1 (6.2)

17. Secondary Outcome: Double Blind Period: Number of Combined Unique Active (CUA) Lesions, Active Time Constant 2 (T2) Lesions, and Time Constant 1 (T1) Gadolinium Enhanced (Gd+) Lesions Per Participant Per Scan
Description: Number of CUA lesions, active T2 lesions, and T1 Gd+ lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: Week 96
Population: ITT population included all randomized participants who had received at least one dose of study medication in the DB period. Here "Number of Participants analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 121 | 48
Lesions
  T1 Gd+ lesions | 0.06 (0.37) | 0.34 (0.87)
  CUA lesions | 0.55 (1.27) | 1.12 (1.94)
  T2 lesions | 0.53 (1.26) | 1.04 (1.81)

18. Secondary Outcome: Double Blind Period: Mean Number of T1 Hypointense Lesions Per Participant Per Scan at Week 96
Description: Mean number of T1 hypointense lesions per participant per scan at 96 weeks were reported. T1 hypointense lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: Week 96
Population: ITT population included all randomized participants who had received at least one dose of study medication in the DB period. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 121 | 48
Lesions | 0.28 (0.63) | 0.43 (1.00)

19. Secondary Outcome: Double Blind Period: Percentage of Participants With no Active T2 Lesions at Week 96
Description: Percentage of participants with no active T2 lesions at week 96 were reported. Active T2 lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: Week 96
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 121 | 48
Percentage of Participants | 56.2 | 29.2

20. Secondary Outcome: Double Blind Period: Percentage of Participants With no Active T1 Gd-Enhanced Lesions at Week 96
Description: Percentage of participants with no active T1 Gd-enhanced lesions at week 96 were reported. Active T1 Gd-Enhanced lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: Week 96
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 121 | 48
Percentage of Participants | 86.0 | 56.3

21. Secondary Outcome: Double Blind Period: Mean Change in T2 Lesion Volume From Baseline to Week 96
Description: Mean change in T2 lesion volume From baseline to Week 96 were reported. T2 lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: Baseline, Week 96
Population: ITT population included all randomized participants who had received at least one dose of study medication in the DB period. Here "Number of participants analyzed" signifies those participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: cubic millimeters (mm^3)
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 105 | 37
cubic millimeters (mm^3) | -2007.2 (3718.3) | -1224.6 (7056.3)

22. Secondary Outcome: Double Blind Period: Percent Change in Normalized Brain Volume From Baseline to Week 96
Description: Brain volume was measured using magnetic resonance imaging (MRI) scans of the brain. Percent change in normalized brain volume from baseline to week 96 was reported.
Time Frame: Baseline, Week 96
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 15 | 6
Percent Change | -1.01 (1.03) | -1.42 (0.73)

23. Secondary Outcome: Double Blind Period: Mean Change in T1 Hypointense Lesion Volume From Baseline to Week 96
Description: Mean change in T1 hypointense lesion volume from baseline to week 96 was reported. T1 Hypointense lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: Baseline, Week 96
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: millimeter cubic
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 105 | 37
millimeter cubic | -481.8 (1097.2) | -263.0 (1678.3)

24. Secondary Outcome: Double Blind Period: Annualized Qualifying Relapse Rate
Description: A qualifying relapse was defined as a 2-grade increase in at least one, or a 1-grade increase in at least two, Kurtzke Functional Systems excluding bowel/bladder or cognition changes, in the absence of fever lasting more than or equal to 24 hours, and preceded by more than or equal to 30 days of clinical stability or improvement. The annualized relapse rate for each treatment group was the mean of the annualized relapse rates for all the participants in the group, calculated as the total number of confirmed relapses divided by the total number of days on study multiplied by 365.25.
Time Frame: Baseline up to Week 96
Population: ITT population included all randomized participants who had received at least one dose of study medication in the DB period.
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 124 | 48
relapses per year | 0.12 [0.08 to 0.17] | 0.32 [0.20 to 0.45]
Statistical Analysis 1: Comparison: Cladribine 3.5 mg/kg, IFN-beta (DB Period) vs Placebo, IFN-beta (DB Period); Test type: Superiority; p < 0.001, Wald Chi-square; Relative Risk = 0.37, 95% CI 2-sided [0.22 to 0.63]

25. Secondary Outcome: Double Blind Period: Percentage of Participants Qualifying Relapse-free
Description: A qualifying relapse was defined as a 2-grade increase in 1 or more Kurtzke Functional Systems (KFS) or a 1-grade increase in 2 or more KFS, excluding changes in bowel/bladder or cognition, in the absence of fever, lasting for >= 24 hours, and preceded by at least 30 days of clinical stability or improvement. Percentage of participants qualifying relapse-free were reported.
Time Frame: Baseline up to Week 96
Population: as for outcome 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 124 | 48
Percentage of Participants | 75.0 | 52.1

26. Secondary Outcome: Double Blind Period and OLE Period: Time to 3-Month Sustained Expanded Disability Status Scale (EDSS) Progression
Description: EDSS progression is based on a standardized neurological exam and focuses on symptoms that commonly occur in Multiple Sclerosis (MS). Overall scores ranges from 0.0 (normal) to 10.0 (death due to MS). A sustained progression on EDSS score was defined as an EDSS progression confirmed into two consecutive assessment. Time to sustained disability progression was analyzed using a Cox proportional hazards model. 10th and 20th percentiles estimated from Kaplan-Meier survival curve. Due to the small number of events, estimates from Kaplan-Meier survival curves could only be derived for lower percentiles. The median (50th percentile) could not be estimated if less than 50% of the participants had an event during the time of the study. Accordingly, lower percentiles are presented according to the number of events observed.
Time Frame: Baseline up to Week 96
Population: ITT population included all randomized participants who had received at least one dose of study medication in the DB period. Here "Number of Participants analyzed"= participants evaluable for this outcome measure and "number analyzed"= participants who were evaluable for specified category.
Measure: Number; unit: Days
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period) | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 19 | 6 | 10 | 5
Days
  10th percentile | 244 | 484 | 87 | 85
  20th percentile | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | 0 | 246 | 0

27. Secondary Outcome: Double Blind Period and OLE Period: Time to First Qualifying Relapse
Description: A qualifying relapse was defined as a 2-grade increase in at least one, or a 1-grade increase in at least two, Kurtzke Functional Systems excluding bowel/bladder or cognition changes, in the absence of fever lasting more than or equal to 24 hours, and preceded by more than or equal to 30 days of clinical stability or improvement. Time to first qualifying relapse were analyzed using a Cox proportional hazards model. 10th and 20th percentiles estimated from Kaplan-Meier survival curve. Due to the small number of events, estimates from Kaplan-Meier survival curves could only be derived for lower percentiles. The median (50th percentile) could not be estimated if less than 50% of the participants had an event during the time of the study. Accordingly, lower percentiles are presented according to the number of events observed.
Time Frame: Baseline up to Week 96
Population: as for outcome 26
Measure: Number; unit: Days
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period) | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 23 | 16 | 4 | 4
Days
  10th percentile | 239 | 252 | 255 | 155
  20th percentile | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | 481 | 0 | 0

28. Primary Outcome: Open Label Extension Period: Maximum Corrected QT Interval (Qtc)
Description: as for outcome 7
Time Frame: Baseline up to Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 47 | 27
Milliseconds | 0.4370 (0.0219) | 0.4317 (0.0181)

29. Primary Outcome: Open Label Extension Period: Mean Change From Baseline in Vital Signs- Systolic and Diastolic Blood Pressure
Description: Mean change from baseline in vital signs- systolic and diastolic blood pressure was reported.
Time Frame: Baseline, Week 72
Population: Safety population was used. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Only those participants with data available at the specified time point were reported.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mm*hg)
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 3 | 0
Millimeter of mercury (mm*hg)
  Systolic Blood Pressure | 0.3 (10.2) |
  Diastolic Blood Pressure | -1.7 (5.0) |

30. Primary Outcome: Open Label Extension Period: Mean Change From Baseline in Vital Signs- Pulse Rate
Description: Mean change from baseline in vital signs- Pulse Rate was reported.
Time Frame: Baseline, Week 72
Population: Safety population: all randomized participants who received at least 1 dose of study drug in DBP and had follow-up safety data. Here "Number of Participants analyzed"= participants evaluable for this outcome measure. Only those participants with data available at the specified time point were reported.
Measure: Mean (Standard Deviation); unit: beats per minutes
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 3 | 0
beats per minutes | 4.7 (11.5) |

31. Primary Outcome: Open Label Extension Period: Mean Change From Baseline in Vital Signs- Weight
Description: Mean change from baseline in vital signs- weight was reported.
Time Frame: Baseline, Week 72
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 3 | 0
Kilogram | -9.4 (6.9) |

32. Primary Outcome: Open Label Extension Period: Mean Change From Baseline in Vital Signs- Temperature
Description: Mean change from baseline in vital signs- temperature was reported.
Time Frame: Baseline, Week 72
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 3 | 0
Degree celsius | -0.3 (0.3) |

33. Primary Outcome: Open Label Extension Period: Mean Change From Baseline in Electrocardiogram (ECG) Parameters- Heart Rate
Description: Mean change from baseline in ECG parameters- Heart Rate was reported.
Time Frame: Baseline, Week 72
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: beats per minutes
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 6 | 0
beats per minutes | -4.889 (6.160) |

34. Primary Outcome: Open Label Extension Period: Mean Change From Baseline in Electrocardiogram (ECG) Parameters- PR, RR, QRS and OT Interval
Description: Mean change from baseline in ECG parameters- PR, RR, QRS and OT interval was reported.
Time Frame: Baseline, Week 72
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 6 | 0
milliseconds
  PR Interval | -0.0044 (0.0108) |
  RR Interval | 0.0643 (0.0721) |
  QRS Interval | -0.0026 (0.0090) |
  QT Interval | 0.0109 (0.0206) |

35. Secondary Outcome: Double Blind Period: Mean Change in New T1 Gd+ Lesions From Baseline to Week 96
Description: Mean change in new T1 Gd+ lesions from baseline to week 96 was reported.
Time Frame: Baseline, Week 96
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period)
Number analyzed (Participants) | 105 | 37
Lesions | -1.0 (4.4) | -0.3 (1.1)

36. Primary Outcome: OLE and Safety Follow-up Period: Percentage of Participants With Grade 3 or 4 (Common Terminology Criteria for Adverse Events [CTCAE] v 4.0) Hematological or Liver Toxicity
Description: as for outcome 1
Time Frame: Baseline (OLEP) up to Week 96
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) | Placebo, IFN-beta (Safety Follow up)
Number analyzed (Participants) | 47 | 28 | 51 | 7
Percentage of participants
  Grade 3 or 4 Lymphocyte toxicity | 48.9 | 28.6 | 3.9 | 0.00
  Grade 3 or 4 Hemoglobin toxicity | 0.00 | 0.00 | 2.0 | 0.00
  Grade 3 or 4 White Blood Cell toxicity | 4.3 | 3.6 | 0.00 | 0.00
  Grade 3 or 4 Neutrophil toxicity | 6.4 | 14.3 | 0.00 | 0.00
  Grade 3 or 4 CD4+ toxicity: number analyzed (Participants) | 47 | 28 | 50 | 7
  Grade 3 or 4 CD4+ toxicity | 66.0 | 21.4 | 14.0 | 0.00
  Grade 3 or 4 AST toxicity | 0.00 | 0.00 | 0.00 | 0.00
  Grade 3 or 4 ALT toxicity | 0.00 | 3.6 | 0.00 | 0.00
  Grade 3 or 4 Platelet toxicity | 0.00 | 0.00 | 0.00 | 0.00
  Grade 3 or 4 Bilirubin toxicity | 0.00 | 0.00 | 0.00 | 0.00

37. Primary Outcome: OLE and Safety Follow-up Period: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) in Infections and Infestations System Organ Class (SOC)
Description: as for outcome 2
Time Frame: Baseline (OLEP) up to Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) | Placebo, IFN-beta (Safety Follow up)
Number analyzed (Participants) | 47 | 28 | 52 | 7
Percentage of participants | 38.3 | 21.4 | 11.5 | 0

38. Primary Outcome: OLE and Safety Follow-up Period: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: as for outcome 3
Time Frame: Baseline (OLEP) up to Week 96
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) | Placebo, IFN-beta (Safety Follow up)
Number analyzed (Participants) | 47 | 28 | 52 | 7
Participants
  Participants with TEAEs | 37 | 19 | 22 | 0
  Participants with Serious TEAEs | 0 | 1 | 1 | 0

39. Primary Outcome: Open Label Extension Period: Time to First Grade 3 or 4 Hematological Toxicity or Liver Toxicity
Description: Time to first Grade 3 or 4 hematological toxicity or liver toxicity (lymphocytes, cluster of differentiation 4 (CD4+) cell, neutrophils, white blood cells, hemoglobin, Alanine transaminase (ALT), Aspartate transaminase (AST), Platelets and Bilirubin) were estimated using the Kaplan-Meier method. According to CTCAE v 4.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death. 10th and 20th percentiles estimated from Kaplan-Meier survival curve. Due to the small number of events, estimates from Kaplan-Meier survival curves could only be derived for lower percentiles. The median (50th percentile) could not be estimated if less than 50% of the participants had an event during the time of the study. Accordingly, lower percentiles are presented according to the number of events observed.
Time Frame: Baseline up to Week 96
Population: as for outcome 4
Measure: Number; unit: Months
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext)
Number analyzed (Participants) | 31 | 8
Months
  10th percentile: Lymphocytes toxicity: number analyzed (Participants) | 23 | 8
  10th percentile: Lymphocytes toxicity | 0.30 | 0.36
  20th percentile: Lymphocytes toxicity: number analyzed (Participants) | 23 | 8
  20th percentile: Lymphocytes toxicity | 1.64 | 2.23
  10th percentile:Hemoglobin toxicity: number analyzed (Participants) | 0 | 0
  20th percentile:Hemoglobin toxicity: number analyzed (Participants) | 0 | 0
  10th percentile: White Blood Cell toxicity: number analyzed (Participants) | 2 | 1
  10th percentile: White Blood Cell toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: White Blood Cell toxicity: number analyzed (Participants) | 2 | 1
  20th percentile: White Blood Cell toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: Neutrophil toxicity: number analyzed (Participants) | 3 | 4
  10th percentile: Neutrophil toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | 0.92
  20th percentile: Neutrophil toxicity: number analyzed (Participants) | 3 | 4
  20th percentile: Neutrophil toxicity | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: Platelets toxicity: number analyzed (Participants) | 0 | 0
  20th percentile: Platelets toxicity: number analyzed (Participants) | 0 | 0
  10th percentile: CD4+ count toxicity: number analyzed (Participants) | 31 | 6
  10th percentile: CD4+ count toxicity | 0.92 | 2.96
  20th percentile: CD4+ count toxicity: number analyzed (Participants) | 31 | 6
  20th percentile: CD4+ count toxicity | 0.99 | 7.00
  10th percentile: AST toxicity: number analyzed (Participants) | 0 | 0
  20th percentile: AST toxicity: number analyzed (Participants) | 0 | 0
  10th percentile: ALT toxicity: number analyzed (Participants) | 0 | 1
  10th percentile: ALT toxicity |  | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: ALT toxicity: number analyzed (Participants) | 0 | 1
  20th percentile: ALT toxicity |  | NA — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: Bilirubin toxicity: number analyzed (Participants) | 0 | 0
  20th percentile: Bilirubin toxicity: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: DB Period: Baseline up to Week 96; OL Extension Period and Safety follow-up period: Baseline up to Week 96
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Cladribine 3.5 mg/kg, IFN-beta (DB Period) | Placebo, IFN-beta (DB Period) | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) | Placebo, IFN-beta (Safety Follow up)
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/48 | 0/47 | 0/28 | 0/52 | 0/7
Serious Adverse Events (participants affected / at risk) | 12/124 | 5/48 | 0/47 | 1/28 | 1/52 | 0/7
Other Adverse Events (participants affected / at risk) | 111/124 | 33/48 | 24/47 | 12/28 | 0/52 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine 3.5 mg/kg, IFN-beta (DB Period) (N=124) | Placebo, IFN-beta (DB Period) (N=48) | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) (N=47) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) (N=28) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) (N=52) | Placebo, IFN-beta (Safety Follow up) (N=7)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Human ehrlichiosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Atonic urinary bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine 3.5 mg/kg, IFN-beta (DB Period) (N=124) | Placebo, IFN-beta (DB Period) (N=48) | Cladribine 3.5 mg/kg, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) (N=47) | Placebo, IFN-beta, Cladribine 3.5 mg/kg (OL Ext) (N=28) | Cladribine 3.5 mg/kg, IFN-beta (Safety Follow up) (N=52) | Placebo, IFN-beta (Safety Follow up) (N=7)
Lymphopenia (Blood and lymphatic system disorders) | 50 | 0 | 11 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 13 | 3 | 3 | 3 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 14 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 18 | 6 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 13 | 4 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 13 | 4 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 7 | 3 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 4 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 28 | 8 | 3 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 8 | 3 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 15 | 6 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 14 | 5 | 1 | 4 | 0 | 0
Influenza (Infections and infestations) | 7 | 4 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 7 | 2 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 7 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 13 | 0 | 4 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 4 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 31 | 10 | 6 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 3 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 3 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 7 | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 3 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 3 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The 96-week DB treatment period of study was completed as planned, and safety and exploratory efficacy results are presented here. The duration of OL Ext. period was reduced for some participants, following termination of the development program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other